CLINICAL TRIAL: NCT00535184
Title: A Multicenter Study to Test Digital Breast Tomosynthesis (DBT) Compared to Full-Field Digital Mammography (FFDM) in Detecting Breast Cancer. Part 3. Women Undergoing Breast Biopsy
Brief Title: Test of Digital Breast Tomosynthesis vs. Common Mammography to Detect Breast Cancer for Women Undergoing Breast Biopsy
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: GE 190-003
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: Mammography; mammogram; breast; Abnormal and normal breast tissue
MeSH Terms: conditions — Breast Neoplasms; Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of the ability of DBT and FFDM to detect breast cancer.

DETAILED DESCRIPTION:
Enrolled women will undergo bilateral DBT. Prior breast imaging data (screening and diagnostic mammography) must have been conducted on GE equipment and the images must be available (or imaging must be repeated). DBT images will be read on-site by one or more qualified radiologists. All subjects who undergo biopsy will be asked to return in approximately 1 year for a follow-up mammogram. Images will be processed and evaluated by independent readers.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years or older and has underwent screening/diagnostic mammography and referred for breast biopsy
* Able and willing to comply with study procedures, and have signed and dated the informed consent form
* Surgically sterile or postmenopausal

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Has signs or symptoms of breast cancer
* Has been previously included in this study
* Has breast implants
* Has a history of breast cancer and is in active treatment
* Has breasts too large to be adequately positioned for the DBT examination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women referrd for breast biopsy because of one or more abnormalities seen on routine screening mammography; who are also asymptomatic
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Longcore, Study Director — GE Healthcare